CLINICAL TRIAL: NCT00448201
Title: Allogeneic Hematopoietic Cell Transplantation for Patients With Hematologic Disorders Who Are Ineligible or Inappropriate for Treatment With a More Intensive Therapeutic Regimen
Brief Title: Reduced-Intensity Busulfan and Fludarabine With or Without Antithymocyte Globulin Followed by Donor Stem Cell Transplant in Treating Patients With Hematologic Cancer or Other Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0306; P30CA016086 (NIH)
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); prolymphocytic leukemia; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; primary myelofibrosis; Waldenstrom macroglobulinemia; adult nasal type extranodal natural killer (NK)/T-cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Prolymphocytic; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Leukemia, Myeloid, Acute; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Primary Myelofibrosis; Waldenstrom Macroglobulinemia; Lymphoma, Extranodal NK-T-Cell | interventions — Antilymphocyte Serum; sargramostim; Busulfan; fludarabine phosphate; Methotrexate; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Methotrexate Only Arm (Active Comparator): GVHD Prophylaxis with Methotrexate
  Interventions: Biological: sargramostim; Biological: therapeutic allogeneic lymphocytes; Drug: busulfan; Drug: fludarabine phosphate; Drug: methotrexate; Drug: tacrolimus; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation
- 2 Doses ATG + Methotrexate (Active Comparator): GVHD prophylaxis with antithymocyte globulin (ATG) + Methotrexate
  Interventions: Biological: anti-thymocyte globulin; Biological: sargramostim; Biological: therapeutic allogeneic lymphocytes; Drug: busulfan; Drug: fludarabine phosphate; Drug: methotrexate; Drug: tacrolimus; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation
- 2 Doses ATG (Active Comparator): GVHD prophylaxis with 2 doses ATG
  Interventions: Biological: anti-thymocyte globulin; Biological: sargramostim; Biological: therapeutic allogeneic lymphocytes; Drug: busulfan; Drug: fludarabine phosphate; Drug: tacrolimus; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation
- 3 Doses ATG (Active Comparator): GVHD prophylaxis with 3 doses ATG
  Interventions: Biological: anti-thymocyte globulin; Biological: sargramostim; Biological: therapeutic allogeneic lymphocytes; Drug: busulfan; Drug: fludarabine phosphate; Drug: tacrolimus; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin — 0.5 mg/kg on day -3, 2.5 mg/kg on day -2 (groups 2, 3 and 4) and 3 mg/kg on day -1 (group 4 only)
  Arms: 2 Doses ATG; 2 Doses ATG + Methotrexate; 3 Doses ATG
Biological: sargramostim — GM-CSF 500 ug everyday (QD) subcutaneously will be given to recipients who remain with an Absolute neutrophil count (ANC) < 1000/microliter (uL) past day 20
Biological: therapeutic allogeneic lymphocytes — A minimum total cluster of differentiation 34 (CD34)+ cell dose of 3 x 10^6 cells/kg and a maximum 8 x 10^6 cells/kg will be infused on day 0
Drug: busulfan — 6.4 mg/kg by continuous IV infusion over 48 hours on Days -6 and -5
Drug: fludarabine phosphate — fludarabine 30 mg/m^2/day x 5 days IV piggyback (IVPB) over 30 minutes on Days -7 through -3
Drug: methotrexate — Methotrexate 5 mg/m^2 per day on days +1, +3 and +6
  Arms: 2 Doses ATG + Methotrexate; Methotrexate Only Arm
Drug: tacrolimus — Suggested starting dose is 0.03 mg/kg po bid starting on Day -1
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Minimum total CD34+ cells of 3 x 10^6 cells/kg and a maximum of 8 x 10^6 cells/kg will be infused on Day 0
Procedure: peripheral blood stem cell transplantation — Minimum total CD34+ cells of 3 x 10^6 cells/kg and a maximum of 8 x 10^6 cells/kg will be infused on Day 0

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as busulfan and fludarabine, before a donor stem cell transplant helps stop the growth of cancer and abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer or abnormal cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Immunosuppressive therapy may improve bone marrow function and may be an effective treatment for hematologic cancer or other disease.

PURPOSE: This clinical trial is studying the side effects and how well giving busulfan and fludarabine with or without antithymocyte globulin followed by donor stem cell transplant works in treating patients with hematologic cancer or other disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical efficacy and toxicity profiles of a nonmyeloablative preparative regimen comprising busulfan and fludarabine with or without anti-thymocyte globulin followed by allogeneic hematopoietic stem cell transplantation in patients with hematologic cancers or other diseases.
* Determine the feasibility of this regimen in these patients.
* Establish a treatment-related mortality during the first 6 months that is less than 20% in patients treated with this regimen.

Secondary

* Determine the response rates (disease-specific partial response and complete response) in patients treated with this regimen.
* Determine overall and progression-free survival of patients treated with this regimen.
* Determine the percent donor chimerism and immunologic recovery, including dendritic cell recovery, in patients treated with this regimen.
* Determine the risk of acute and chronic graft-versus-host disease and other toxicities in patients treated with this regimen.
* Assess the overall nonhematologic grades 3 and 4 toxicity of this regimen, including the incidence of veno-occlusive disease and pulmonary toxicity, in these patients.

OUTLINE: Patients are assigned to 1 of 4 treatment groups according to disease type and donor type.

* Preparative regimen:

  * Group 1 (patients with acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), IPSS (International Prognostic Scoring System score) high-risk myelodysplastic syndromes (HR MDS), or chronic myelogenous leukemia (CML) with an human leukocyte antigen (HLA)-matched related donor (MRD): Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -3 and busulfan IV continuously over 48 hours on days -6 and -5.
  * Group 2 (patients with AML, ALL, IPSS HR MDS, or CML with an HLA-matched unrelated donor (MUD) or mismatched related donor (MMRD)): Patients receive fludarabine phosphate and busulfan as in group 1 and anti-thymocyte globulin IV over 4 hours on day -8.
  * Group 3 (patients with all other diseases with a MRD): Patients receive fludarabine phosphate and busulfan as in group 1 and anti-thymocyte globulin as in group 2.
  * Group 4 (patients with all other disease with a MUD or MMRD): Patients receive fludarabine phosphate and busulfan as in group 1 and anti-thymocyte globulin IV over 4 hours on days -8 and -7.
* Allogeneic stem cell transplantation: All patients undergo allogeneic peripheral blood stem cell transplantation on day 0. Patients then receive sargramostim (GM-CSF) subcutaneously once daily beginning on day 5 (groups 1 and 2) or day 7 (groups 3 and 4) and continuing until blood counts recover.
* Graft-vs-host disease (GVHD) prophylaxis: All patients receive oral tacrolimus twice daily on days -1 to 120 followed by a taper until day 180. Patients in groups 1 and 2 also receive methotrexate IV on days 1, 3, and 6.
* Donor lymphocyte infusion (DLI): After day 120, patients with progressive disease or stable disease while off immunosuppression and with no evidence of active GVHD may receive DLI. Treatment with DLI may repeat every 8 weeks for up to 3 total infusions in the absence of disease response or GVHD.

Peripheral blood and/or bone marrow samples are collected at baseline and then at 30, 60, 90, 120, and 180 days post-transplantation. Chimerism (including the following subsets: whole blood, T-cells as defined by cluster of differentiation 3 (CD3) positivity, B-cells as defined by Cluster of Differentiation 19 (CD19) positivity, and myeloid cells as defined by Cluster of Differentiation 14 (CD14) and Cluster of Differentiation 15 (CD15) positivity is analyzed by polymerase chain reaction technology.

After restaging between Days 90 and 100 and between Days 150 to 180, patients are followed every 6 months for 1 years and then yearly for a maximum of 5 years from study entry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Chronic lymphocytic leukemia (CLL), meeting the following criteria:

    * Absolute lymphocyte count > 5,000/mm³
    * Lymphocytes must appear morphologically mature with < 55% prolymphocytes
    * Lymphocyte phenotype with expression of CD19 and cluster of differentiation 5 (CD5)
  * Prolymphocytic leukemia (PLL), meeting the following criteria:

    * Absolute lymphocyte count > 5,000/mm³
    * More than 55% prolymphocytes
    * Morphologically diagnosed
  * Chronic myelogenous leukemia (CML), meeting the following criteria:

    * Diagnosis of CML or similar myeloproliferative disorders based on t(9;22) or related t(9;12) cytogenetic abnormalities AND characterized by elevated white blood cell (WBC) counts in peripheral blood or bone marrow
    * In first chronic phase CML and a candidate for treatment with reduced-dose busulfan
    * Patients with other cytogenetic abnormalities, such as t(9;12), that are associated with an aggressive clinical course are eligible
  * Non-Hodgkin's lymphoma (NHL), meeting the following criteria:

    * Any World Health Organization (WHO) class histologic subtype allowed
    * Core biopsies are acceptable provided they contain adequate tissue for primary diagnosis and immunophenotyping
    * Bone marrow biopsies as sole means of diagnosis are not allowed for follicular lymphoma
  * Hodgkin's lymphoma, meeting the following criteria:

    * Any WHO class histologic subtype allowed
    * Core biopsies are acceptable provided they contain adequate tissue for primary diagnosis and immunophenotyping
  * Multiple myeloma, meeting the following criteria:

    * Active disease requiring treatment (Durie-Salmon stages I, II, or III)
  * Acute myeloid leukemia with documented control, defined as < 10% bone marrow blasts and no circulating blasts
  * Acute lymphoblastic leukemia, meeting the following criteria:

    * In early first relapse or beyond OR in first complete remission and has 1 of the following high-risk features:

      * t(9;22) or t(4;11)
      * WBC count > 30,000/mm³ at presentation
      * Non-T-cell phenotype
      * More than 30 years of age
  * Agnogenic myeloid metaplasia/myelofibrosis

    * Patients who are transfusion dependent or who have evolving myelodysplastic or leukemic features or high-risk cytogenetic abnormalities are eligible
  * Myelodysplastic syndromes (MDS) as defined by WHO criteria
* Meets 1 of the following criteria:

  * Over 55 years of age
  * Ineligible for busulfan-based therapy based on diminished organ function or poor performance status
  * Indolent and chemotherapy-responsive CLL, low-grade NHL, small lymphocytic lymphoma, or PLL
* Patients who have undergone prior autologous stem cell transplantation are preferentially enrolled on clinical trial CALGB-100002, if available and patient is eligible
* HLA-matched or mismatched related donor or HLA-matched unrelated donor available

  * HLA-identical sibling (6/6 or 9/10) (minimal serologic typing required for class I [A, B]; molecular typing required for class II (DRB1))
  * 9/10 matched unrelated donor (MUD) (molecular analysis at HLA A, B, C, DRB1, and DQB1 by high resolution typing required)
  * 5/6 MUD (molecular analysis at HLA A, B, and DRB1 required)
  * No syngeneic donors

PATIENT CHARACTERISTICS:

* Creatinine clearance ≥ 40 mL/min
* Bilirubin ≤ 3 times upper limit of normal (ULN)
* aspartate aminotransferase (AST) ≤ 3 times ULN
* Diffusing capacity of the lungs for carbon monoxide (DLCO) > 40% with no symptomatic pulmonary disease
* Left ventricular ejection fraction (LVEF) ≥ 30% by multigated acquisition scan (MUGA)
* No uncontrolled diabetes mellitus or active serious infection
* No known hypersensitivity to Escherichia coli-derived products
* No HIV infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy, radiotherapy (except prophylactic cranial x-ray therapy), or surgery

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-01-07 (Actual); Primary Completion 2011-01-11 (Actual); Study Completion 2012-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Shea, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina (UNC) Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with histologically confirmed hematologic malignancies, who were over the age of 55, or otherwise ineligible for more intensive busulfan-based therapy were enrolled on protocol Lineberger Comprehensive Cancer Center (LCCC) 0306 at the University of North Carolina.
Groups:
- All Trial Participants: All patients received IV fludarabine 30 mg/m2/day on days -7 through -3; busulfan 6.4 mg/kg by continuous infusion over 48 hours on days -6 through -5 and tacrolimus from day -1. Throughout the study duration, 8 different GVHD regimens were investigated. In addition to tacrolimus, patients received combinations of 3 agents: methotrexate (5 mg/m2 D1, 3, 6), rabbit antithymocyte globulin (ATG, 3 mg/kg to- 6 mg/kg) or alemtuzumab (Campath, 30 mg to- 90 mg).
Period: Overall Study
Arm/Group | All Trial Participants
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Trial Participants
Number analyzed (Participants) | 71
Age, Continuous [Median (Full Range); unit: years] | 58 [28 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 60
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 71
Donor Types [Count of Participants; unit: Participants] — Human leukocyte antigen (HLA) typing is used to match a recipient with a donor for bone marrow or cord blood transplant. Donor types are either HLA-matched related donor (MRD) or matched unrelated donor (MUD) or HLA-mismatched grafts.
  Participants
    HLA-matched related donor (MRD) | 37
    MUD or HLA-mismatched grafts | 34
Comorbidity Index (CI) [Median (Full Range); unit: units on a scale] — The Hematopoietic Cell Transplantation-Specific Comorbidity Index (HCT-CI) was developed to identify relevant comorbidities in the allogeneic stem cell transplantation population and to enable risk assessment before allogeneic transplant. Comorbidities are given a a weighted score of 1 to 3 if present. The total score can range from 0 to 29, with higher numbers indicating more/worse comorbidities. The HCT-CI scores were further collapsed into 3 risk groups: 0 (low risk), 1 to 2 (intermediate risk), and 3 or more (high risk).
  units on a scale | 3 [0 to 8]
Disease Risk Index (DRI) [Count of Participants; unit: Participants] — The DRI uses a combination of a ternary breakdown for disease type and a binary breakdown for remission status to assign patients to 1 of 4 risk categories that differ very significantly (statistically and clinically) with respect to overall survival (OS) and Progression free survival (PFS).
  Participants
    Low | 9
    Intermediate | 40
    High | 19
    Very High | 1
    Undetermined | 2

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Mortality
Description: Treatment related mortality for first 6 months. Defined as the number of treatment related deaths excluding deaths due to disease relapse.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | All Trial Participants
Number analyzed (Participants) | 71
percentage of participants | 8.4

2. Secondary Outcome: Complete Response at 6 and 12 Months Post-transplant
Time Frame: 6 and 12 months
Population: Complete response was not calculated at 6 and 12 months because the majority of patients had complete response at the time of transplant.
Arm/Group | All Trial Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Complete or Mixed Donor Chimerism at 30, 60, and 90 Days Post-transplant
Description: Complete chimerism is defined as 100% donor cells detected, suggesting complete hematopoietic replacement. Mixed donor chimerism means host cells are detected in particular cells like lymphocytes. Five to 90% donor cells set the criteria for mixed chimerism (MC).
  Chimerism was not tabulated on day 30.
Time Frame: Days 30, 60, and 90
Measure: Number; unit: percentage of patients
Groups:
- Day 60: 60 days post-transplant
- Day 90: 90 days post-transplant
Arm/Group | Day 60 | Day 90
Number analyzed (Participants) | 71 | 71
percentage of patients
  Complete Donor | 82 | 87
  Mixed Donor | 18 | 13

4. Secondary Outcome: 5-year Disease-free Survival
Description: The length of time post-transplant that the patient survives without any signs or symptoms of that cancer.
Time Frame: Year 5
Measure: Number; unit: percentage of participants
Arm/Group | All Trial Participants
Number analyzed (Participants) | 71
percentage of participants | 31

5. Secondary Outcome: Graft-vs-host Disease at 6 Months Post-transplant
Description: Graft-vs-host disease (GVHD) can be mild, moderate or severe depending on the differences in tissue type between patient and donor. Its symptoms can include:
  * Rashes, which include burning and redness, that erupt on the palms or soles and may spread to the trunk and eventually to the entire body
  * Blistering, causing the exposed skin surface to flake off in severe cases
  * Nausea, vomiting, abdominal cramps, diarrhea and loss of appetite, which can indicate that the gastrointestinal (digestive) tract is affected
  * Jaundice, or a yellowing of the skin, which can indicate liver damage
  * Excessive dryness of the mouth and throat, leading to ulcers
  * Dryness of the lungs, vagina and other surfaces
  Acute GVHD - Can occur soon after the transplanted cells begin to appear in the recipient. Acute GVHD ranges from mild, moderate or severe, and can be life-threatening if its effects are not controlled.
  Extensive chronic GVHD - Usually occurs at about three months post-transplant.
Time Frame: 6 Months
Measure: Number; unit: percentage of participants
Arm/Group | All Trial Participants
Number analyzed (Participants) | 71
percentage of participants
  Acute GVHD | 13
  Extensive Chronic GVHD | 30

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | All Trial Participants
All-Cause Mortality (participants affected / at risk) | 44/71
Serious Adverse Events (participants affected / at risk) | 7/71
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Trial Participants (N=71)
hypoxemia (Blood and lymphatic system disorders) | 1
graft failure (Blood and lymphatic system disorders) | 1
liver toxicity/hyperbilirubinemia (Hepatobiliary disorders) | 1
Graft vs host disease grade 4 (Gastrointestinal disorders) | 3
CMV viremia (Infections and infestations) | 1
subdural hematoma (Vascular disorders) | 1
Fever (Infections and infestations) | 2
Failure to thrive (General disorders) | 1
elevated lipase (Gastrointestinal disorders) | 1
CMV pneumonia (Infections and infestations) | 1
BK viruria (Infections and infestations) | 1
fungal pneumonia (Infections and infestations) | 1
bronchiolitis obliterans organizing pneumonia (Infections and infestations) | 1
EBV viremia (Infections and infestations) | 1
nocardia pneumonia (Infections and infestations) | 1
toxic epidermal nectrolysis (General disorders) | 1

LIMITATIONS AND CAVEATS:
Per the protocol, non-serious adverse events were not captured as this was a high-dose transplant study and grades 1,2, and 3 adverse events were expected. No unexpected toxicities were seen beyond those reported in the Serious Adverse Event section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes